CLINICAL TRIAL: NCT02289105
Title: The Impact of Active Choice on Completion Rates of Advanced Directives in New Employees of an Academic University Hospital
Brief Title: Impact of Active Choice on Advance Directive Completion Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 818456
Record Dates: First submitted 2014-11-05; First posted 2014-11-13 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Advance Directive Completion
Keywords: Advance Directive; Active Choice; Decision making

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mandatory active choice (Experimental): The mandatory active choice group will be presented two forms at the same time. The first form will be a legally valid AD. The second form will be a declination form. Participants in the intervention arm will be required to complete, and submit either of the two forms the task.
  Interventions: Behavioral: Mandatory active choice
- Control (No Intervention): Participants in the control group will be presented an AD form only and will be encouraged to complete, and submit the form without having to declare the choice of completing or declining the AD.

INTERVENTIONS:
Behavioral: Mandatory active choice — the mandatory active choice group, will be presented two forms at the same time. The first form will be a legally valid AD. The second form will be a declination form. Participants in the intervention arm will be required to complete, and submit either of the two forms the task.
  Arms: Mandatory active choice

SUMMARY:
The overall objective of this project is to assess if an active choice intervention can increase advance directive completion rates.

DETAILED DESCRIPTION:
Nearly 70% of Americans express the desire to die at home, and most individuals want to avoid aggressive or futile care. Despite this, more than half of Americans die in a hospital. Advance directives provide the opportunity to provide, in advance, one's wishes for end of life care, however their completion rates are low. The overall objective of this project is to assess if an active choice intervention can increase AD completion rates. Eligible participants for this study will be all new employees of the University of Pennsylvania Health System (UPHS) who need to complete their online employment paperwork via the On Boarding portal. Participants will have an advanced health care planning task programmed as part of their On Boarding online employment paperwork. Upon selection of the task, each participant will be directed a designated Advance Healthcare Planning (AHCP) website. Participants will be randomized into either the active choice or control arm of the study and proceed through steps to complete or not complete an AD according to the decision making process of the given study arm. All participants in both groups will have access to additional online and telephone resources thought the entire study for any questions. Participants in the active choice group will be given directions stating they are required to complete either the advanced directive or the declination form in order to complete their On Boarding process. Participants in the control group will be given directions stating that completion of the AD is optional.

ELIGIBILITY:
Inclusion Criteria:

* New participants of the University of Pennsylvania Health System who have not yet completed their On Boarding process.
* 18 years of age or older
* Have proficiency in reading, writing, and speaking English

Exclusion Criteria:

* All new UPHS employees will be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1279 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, MD, PhD,, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mandatory Active Choice: The mandatory active choice group could choose to: complete an AD, confirm prior completion of an AD, or complete a form declining AD completion and indicate their reason(s) for doing so.
  Mandatory active choice: the mandatory active choice group, unlike the control group, could not simply skip the task. If they didn't want to complete an AD, they had to fill out a declination form.
- Control: Participants in the control group could choose to: complete an AD, confirm prior AD completion, or skip the task.
Period: Overall Study
Arm/Group | Mandatory Active Choice | Control
Started | 642 | 637
Completed | 642 | 637
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mandatory Active Choice | Control | Total
Number analyzed (Participants) | 642 | 637 | 1279
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [25 to 39] | 29 [25 to 37] | 29 [25 to 38]
Sex/Gender, Customized [Number; unit: participants]
  Male | 446 | 472 | 918
  Female | 186 | 147 | 333
  Prefer not to answer or missing | 10 | 18 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 333 | 345 | 678
  Black | 177 | 167 | 344
  Asian | 51 | 41 | 92
  Mixed or Other | 55 | 50 | 105
  Prefer not to answer or missing | 26 | 34 | 60
Region of Enrollment [Number; unit: participants]
  United States | 642 | 637 | 1279
Employment Status [Number; unit: participants]
  Full-time | 464 | 469 | 933
  Part-time | 178 | 168 | 346
Highest level of education [Number; unit: participants]
  Graduate Degree | 115 | 109 | 224
  College Degree | 304 | 298 | 602
  Some College | 136 | 133 | 269
  High School or Less | 57 | 51 | 108
  Missing | 30 | 46 | 76
Clinical Degree [Number; unit: participants]
  No | 500 | 510 | 1010
  Yes | 142 | 127 | 269

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants That Select to Complete an Advance Directive
Description: We will analyze the effects of the active choice intervention on rates of completion.
Time Frame: Baseline - up to 1 year
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Mandatory Active Choice | Control
Number analyzed (Participants) | 642 | 637
proportion of participants | 0.35 [0.31 to 0.39] | 0.20 [0.17 to 0.24]

2. Secondary Outcome: Proportion of Participants Who Already Have ADs
Time Frame: Baseline - up to 1 year
Measure: Number; unit: proportion of participants
Arm/Group | Mandatory Active Choice | Control
Number analyzed (Participants) | 642 | 637
proportion of participants | .065 | .063

3. Secondary Outcome: Proportion of Participants Who Return a Signed AD
Description: This measures the proportion of participants who return a signed and printed copy of their AD of those who completed an AD online.
Time Frame: Baseline - up to 1 year
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Mandatory Active Choice | Control
Number analyzed (Participants) | 642 | 637
proportion of participants | .078 [.058 to .101] | .039 [.026 to .057]

4. Other Pre Specified Outcome: Participant Selections on ADs and Declination Forms
Time Frame: Baseline - up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: We did not collect or assess serious adverse events because the study is minimal risk.
Arm/Group | Mandatory Active Choice | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/642 | 0/637

LIMITATIONS AND CAVEATS:
Study population is not ideal - healthy workers may not benefit from AD completion as much as older or seriously ill patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No